CLINICAL TRIAL: NCT02744729
Title: Safety and Diagnostic Performance of 99mTc-3PRGD2 SPECT/CT in Esophagus Cancer Patients
Brief Title: 99mTc-3PRGD2 SPECT/CT in Esophagus Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, PhD, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian
Record Dates: First submitted 2016-03-08; First posted 2016-04-20 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esophagus Cancer, 99mTc-3PRGD2, SPECT/CT (Experimental): Determine if 99mTc-3PRGD2 SPECT/CT is safe and effective in diagnosis of Esophagus cancer patients.
  Interventions: Drug: 99mTc-3PRGD2

INTERVENTIONS:
Drug: 99mTc-3PRGD2 — For patients in suspicion of esophagus cancer, single intravenous bolus injection of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 on day one of the treatment period, whole-body planar and thoracic SPECT/CT to determine the accumulation of 99mTc-3PRGD2 in the tumors and the other parts of the body.
  Other Names: 99mTc-HYNIC-3PRGD2

SUMMARY:
This is an open-label single photon emission computed tomography / computed tomography (SPECT/CT) study to investigate the safety and diagnostic performance of 99mTc-HYNIC-3PEG4-E[c(RGDfK)2) (99mTc-3PRGD2) in esophagus cancer patients. A single dose of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the patients in suspicion of esophagus cancer. Visual and semiquantitative method will be used to assess the whole-body planar and thoracic SPECT/CT images. Any adverse events will be collected from the patients.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of integrin receptor family and expressed preferentially on the activated endothelial cells of angiogenesis and some types of tumor cells, but not or very low on the quiescent vessel cells and other normal cells. Therefore, the integrin αvβ3 receptor is becoming a valuable target for diagnosis and response evaluation of malignant tumors.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 expression via single photon emission computed tomography (SPECT)or positron emission tomography (PET). Among all the RGD radiotracers studied, several RGD monomers have been investigated in clinical trials, and the preliminary results demonstrated specific imaging of various types of tumors, and the tumor uptake correlated well with the level of integrin αvβ3 expression. Recently, several RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 99mTc-3PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in animal models to date.

For the further interests in clinical translation of 99mTc-3PRGD2, an open-label SPECT/CT study was designed to investigate the safety and diagnostic performance of 99mTc-3PRGD2 in esophagus cancer patients. A single dose of nearly 11.1 MBq/kg body weight 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the esophagus cancer patients. Visual and semiquantitative method will be used to assess the whole-body planar and thoracic SPECT/CT images. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥30 years old
* Thoracic CT and/or gastroscopy diagnosis in suspicion of primary or recurrent lung cancer.
* The lung cancer will be histologically confirmed or results of histology will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Visual Assessment of Esophagus Lesions in 99mTc-3PRGD2 SPECT/CT Scan | one year
  Visual analysis will be performed by 3 experienced nuclear medicine physicians to observe the the uptake of 99mTc-3PRGD2 on esophagus lesions. The visual analysis interpreter's degree of suspicion for an abnormality was recorded with use of a 3-point with the following categories: score 1, no abnormal increased uptake; score 2, mildly increased uptake; score 3, definite focal increased uptake. The lesion was considered positive as malignancy if the lesion scored as 2 or higher.
Semiquantitative Assessment of Esophagus Lesions in 99mTc-3PRGD2 SPECT/CT Scan | one year
  The semiquantitative analysis of the standardized uptake values (SUV) of 99mTc-3PRGD2 SPECT/CT was performed on esophagus lesion

SECONDARY OUTCOMES:
18F-FDG PET/CT Scan | one year
  18F-FDG PET/CT will be carried out in esophagus cancer patients to assess the uptake of esophagus lesions or distant metastasis and the standardized uptake values (SUVs) of these lesions will be measured.
Laboratory Values | one year
  The blood level of CEA(carcino-embryonic antigen,ng/ml)in participants will be recorded.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of the patients will be followed and assessed. The number of participants with adverse events and abnormal laboratory values will be recorded.
Contrast-enhanced CT | one year
  Contrast-enhanced CT will be carried out in esophagus cancer patients to observe the location and tumor diameter (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes